CLINICAL TRIAL: NCT04506151
Title: Sleep Optimization to Improve Glycemic Control in Adults With Type 1 Diabetes
Acronym: SOPT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Pamela Martyn-Nemeth, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-0374; 1R01DK121726 (NIH)
Record Dates: First submitted 2020-07-22; First posted 2020-08-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Sleep optimization intervention will be compared to an attention control group
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep-Opt (Experimental): 12-week intervention that includes self-monitoring, goal setting, motivational enhancement.
  Interventions: Behavioral: Sleep-Opt
- Healthy Living (Active Comparator): 12-week intervention that includes weekly telephone contact, didactic content equal in time and attention to intervention group.
  Interventions: Behavioral: Healthy Living

INTERVENTIONS:
Behavioral: Sleep-Opt — 12-week behavioral intervention
  Arms: Sleep-Opt
Behavioral: Healthy Living — Healthy Living
  Arms: Healthy Living

SUMMARY:
Up to 40% of adults with type 1 diabetes have insufficient sleep which is associated with negative health consequences including poor blood glucose control and greater diabetes complications. In this study, a sleep intervention (Sleep-Opt) that uses wearable sleep tracking technology, telephone coaching and informational content designed to improve sleep and glycemic control in working-age adults with type 1 diabetes. Sleep-Opt could lead to reduced development of diabetes complications and improve quality of life for adults with type 1 diabetes.

DETAILED DESCRIPTION:
Despite improvements in treatment regimens and technology, less than 20% of adults with type 1 diabetes (T1D) achieve glycemic targets. Sleep is increasingly recognized as a potentially modifiable target for improving glycemic control. Diabetes distress, poor self-management behaviors, and reduced quality of life (QoL) have also been linked to sleep variability and insufficient sleep duration. The American Diabetes Association Standards of Medical Care in Diabetes incorporated sleep as an important component of the medical evaluation in persons with diabetes. However, no specific recommendation was given as to how to improve sleep. A significant gap of knowledge exists regarding the effects of sleep optimization on glycemic control in T1D. The purpose of this study is to determine the efficacy of a T1D-specific sleep optimization intervention (Sleep-Opt) on the primary outcomes of sleep variability, sleep duration and glycemic control (A1C); other glycemic parameters (glycemic variability, time in range), diabetes distress, self-management behavior, QoL, and other patient reported outcomes in working-age adults with T1D and habitual increased sleep variability or short sleep duration. To achieve these aims, a randomized controlled trial is planned in 120 working age adults (18 to 65 years) with T1D. Participants will be screened for habitual sleep variability (> 1 hour/week) or insufficient sleep duration (< 6.5 hours per night). Eligible subjects will be randomized to the Sleep-Opt group or healthy living attention control group for twelve weeks. A one-week run-in period is planned, with baseline measures of sleep by actigraphy (sleep variability and duration), glycemia (A1C and related glycemic measures: glycemic variability and time in range using continuous glucose monitoring), and other secondary outcomes: diabetes distress, self-management behaviors, quality of life and additional patient-reported outcomes. Sleep-Opt is a technology-assisted behavioral sleep intervention that this study team developed that leverages the rapidly increasing public interest in sleep tracking by consumers (+500% in 3 years). The behavioral intervention employs four elements: a wearable sleep tracker, didactic content, an interactive smartphone application, and brief telephone counseling. The attention control group will participate in a healthy living information program. At midpoint (Week 6) completion (Week 12) and post-program (Week 24), baseline measures will be repeated to determine differences between the two groups and sustainability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-65 years
* clinical diagnosis of type 1 diabetes minimum of one year
* reported habitual sleep variability (1 hour/week or more) or sleep duration less than 6.5 hrs/night during work- or weekdays (confirmed with actigraphy sleep watch)
* a desire to improve sleep
* own a smartphone

Exclusion Criteria:

* insomnia symptoms
* at high risk for obstructive sleep apnea
* severe hypoglycemia episode in the past 6 months (e.g. loss of consciousness)
* A1C greater than 10%
* rotating shift or night shift work
* use of sleep medications/aids
* renal impairment (estimated glomerular filtration rate < 45 ml/min)
* significant current medical morbidities (such as heart failure, cirrhosis, chronic obstructive pulmonary disease requiring oxygen, active treatment for cancer, depression, history of stroke with neurological deficits
* breast feeding, pregnant, or planning pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Sleep variability | Change from week 0, 6, 12, 24
  Standard deviation total sleep time for one week
Sleep duration | Change from weeks 0. 6, 12, 24
  total sleep time
Glycemic control | Change from week 0. 6, 12, 24
  HbA1c blood test

SECONDARY OUTCOMES:
Diabetes distress | Change from week 0. 6, 12, 24
  T1D Diabetes Distress Scale score- higher numbers indicate greater distress
Self-management behavior | Change from week. 6, 12, 24
  Self-Management Questionnaire score- higher numbers indicate better self-management
Fatigue | Change from week 0. 6, 12, 24
  Patient Reported Outcomes Measure (PROMIS) fatigue scale score - higher numbers greater fatigue
Mood | Change from week 0. 6, 12, 24
  Center for Epidemiological Studies - Depressed Mood score - Higher numbers more depressive mood

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Martyn-Nemeth, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martyn-Nemeth P, Duffecy J, Quinn L, Reutrakul S, Steffen AD, Burke L, Clark Withington MH, Irsheed GA, Perez R, Park M, Saleh A, Mihailescu D, Baron KG. Sleep optimization to improve glycemic control in adults with type 1 diabetes: study protocol for a randomized controlled parallel intervention trial. Trials. 2022 Aug 19;23(1):686. doi: 10.1186/s13063-022-06565-6. PMID 35986415

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT04506151/Prot_SAP_001.pdf
  • Informed Consent Form (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT04506151/ICF_000.pdf